CLINICAL TRIAL: NCT06173362
Title: A Pragmatic Phase II Study Evaluating Tolerability in Prostate Cancer Patients Treated With Abiraterone + Prednisone or Darolutamide
Brief Title: Abiraterone and Prednisone or Darolutamide for the Treatment of Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mamta Parikh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mamta Parikh, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC315; NCI-2023-09814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC315 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Advanced Prostate Adenocarcinoma; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Specimen Handling; darolutamide; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (abiraterone, prednisone) (Experimental): Patients receive abiraterone and prednisone per SOC. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples during screening and on study.
  Interventions: Drug: Abiraterone; Procedure: Biospecimen Collection; Drug: Prednisone
- Arm II (darolutamide) (Experimental): Patients receive darolutamide per SOC. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Darolutamide

INTERVENTIONS:
Drug: Abiraterone — Given abiraterone
  Other Names: CB 7598
  Arms: Arm I (abiraterone, prednisone)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Darolutamide — Given darolutamide
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201
  Arms: Arm II (darolutamide)
Drug: Prednisone — Given prednisone
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm I (abiraterone, prednisone)

SUMMARY:
This phase II trial compares the effects, good and/or bad of abiraterone and prednisone or darolutamide alone in treating patients with prostate cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Androgens (male hormones) can cause the growth of prostate tumor cells. Abiraterone acetate lowers the amount of androgens made by the body. This may help stop the growth of prostate tumor cells that need androgen to grow. Darolutamide blocks the use of androgens by the tumor cells. Prednisone is used to lessen inflammation and lower the body's immune response. Researchers want to compare the side effects of standard of care (SOC) abiraterone and prednisone or darolutamide alone in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Tolerability.

SECONDARY OBJECTIVES:

I. Tolerability in prespecified subpopulations.

II. Prostate-specific antigen (PSA) response at 7 months.

OUTLINE: Patients are assigned to 1 of 2 arms per treating physician preference.

ARM I: Patients receive abiraterone and prednisone per SOC. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples during screening and on study.

ARM II: Patients receive darolutamide per SOC. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples during screening and on study.

After completion of study intervention, patients are followed up for a total of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an informed consent form
* Histologically confirmed prostate adenocarcinoma
* Advanced prostate cancer appropriate for treatment with abiraterone acetate plus prednisone or darolutamide as assessed by the treating physician
* Participants are encouraged to be currently treated with androgen deprivation therapy (ADT) or having undergone bilateral orchiectomy
* Performance status 0 - 2 (Karnofsky ≥ 50%)
* Age ≥ 18 years at time of consent
* Life expectancy ≥ 6 months per investigator discretion
* Ability and stated willingness to adhere to the study visit schedule and other protocol procedures/requirements for the duration of the study

Exclusion Criteria:

* Have been on either abiraterone or darolutamide for > 28 days prior to initiating enrollment
* Any condition that in the opinion of the investigator would prohibit the understanding or rendering of informed consent or interfere with the participant's safety or compliance while on trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher adverse events | At 12 months
  Will be defined and graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States